CLINICAL TRIAL: NCT00075738
Title: Phase II Study Of 5FU-Irinotecan-Cisplatin As First-Line Treatment In Patients With Metastatic Carcinoma Of The Esophagus
Brief Title: Fluorouracil, Irinotecan, Leucovorin, and Cisplatin as First-Line Therapy in Treating Patients With Metastatic Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000349275; FRE-GERCOR-D00-2; EU-20328
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2007-07

CONDITIONS: Esophageal Cancer
Keywords: stage IV esophageal cancer; recurrent esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cisplatin; Fluorouracil; Irinotecan; Leucovorin

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, irinotecan, leucovorin, and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one chemotherapy drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy as first-line therapy works in treating patients with metastatic esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with metastatic esophageal cancer treated with fluorouracil, irinotecan, leucovorin calcium, and cisplatin as first-line therapy.

Secondary

* Determine the clinical benefit in patients treated with this regimen.
* Determine the tolerability of this regimen in these patients.
* Determine local relapse-free survival of patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive irinotecan IV over 90 minutes and leucovorin calcium IV over 2 hours on day 1. Patients also receive fluorouracil IV continuously over 46 hours and cisplatin IV over 30 minutes on days 1 and 2. Treatment repeats every 15 days for up to 12 courses in the absence of unacceptable toxicity or disease progression.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed esophageal cancer

  * Metastatic disease
* At least 1 unidimensionally measurable metastatic lesion

  * At least 10 mm by spiral scanner OR 20 mm by sequential scanner
  * Outside the field of prior radiotherapy
* No known symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3

Hepatic

* Bilirubin ≤ 1.5 times normal
* Alkaline phosphatase ≤ 3 times normal (5 times normal if liver metastases are present)
* SGOT and SGPT ≤ 3 times normal

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months
* No uncontrolled angina

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy except curatively treated basal cell skin cancer or carcinoma in situ of the cervix
* No other illness or medical condition that would preclude study participation
* No psychological, social, familial, or geographical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 6 months since prior fluorouracil and/or cisplatin
* No other prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 6 weeks since prior radiotherapy

Surgery

* More than 4 weeks since prior surgery

Other

* No concurrent participation in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10

PRIMARY OUTCOMES:
Objective response rate

SECONDARY OUTCOMES:
Clinical benefit
Tolerability
Local relapse-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Artru, MD — Clinique Saint Jean
Locations (15):
- France (15):
  - Clinique La Casamance, Abugne
  - Hopital Saint Andre, Bordeaux
  - Hopital Drevon, Dijon
  - Centre Jean Bernard, Le Mans
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Clinique Saint Jean, Lyon
  - Hopital Notre-Dame de Bon Secours, Metz
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Hopital Haut Leveque, Pessac
  - Clinique Ste - Marie, Pontoise
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Clinique Francois, Saint-Dizier
  - Centre Medico-Chirurgical Foch, Suresnes